CLINICAL TRIAL: NCT01435889
Title: Long Term (1 Year) Respiratory Sequelae in Children Surviving Acute Respiratory Distress Syndrome
Brief Title: Long Term (1 Year) Respiratory Sequelae in Children Surviving an Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: PHRC 2005/R-1906; PHRC 2005/R-1906 (Other Grant/Funding Number: French Ministry of Health)
Record Dates: First submitted 2011-09-16; First posted 2011-09-19 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute respiratory distress syndrome; Children; Long term respiratory sequelae; Pulmonary function tests; Computed tomography, lung
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess long term (1 year) respiratory sequelae in children surviving an acute respiratory distress syndrome

DETAILED DESCRIPTION:
The acute respiratory distress syndrome (ARDS) has a high mortality rate in children. Adverse long term sequelae, and in particular respiratory sequelae, have been described mainly in adults. Decrease in diffusing capacity, lung volume and exercise tolerance were observed. Lung function parameters improve during the follow-up until 6 month after discharge from the pediatric intensive care unit (PICU). After that, abnormalities in PFT are observed in a significant proportion of patients. Only two studies described long-term sequelae in children surviving to an ARDS and their results are conflicting. Two studies carried out in adults described the morphologic long-term sequelae by thoracic computed tomography. They showed reticular pattern with a striking anterior distribution in most patients evaluated more than 6 months after discharge from the PICU. There is, to our knowledge, no study describing morphologic pulmonary sequelae by thoracic computed tomography in children surviving to ARDS.

Respiratory assessment: respiratory sequelae in children surviving to the acute respiratory distress syndrome will be evaluated 1 year after discharge from the PICU. Assessment will include a clinical evaluation (respiratory history and physical examination), respiratory function tests and thoracic computed tomography

ELIGIBILITY:
Inclusion Criteria:

* children surviving to an acute respiratory distress syndrome and alive 1 year after discharge from the PICU

Exclusion Criteria:

* children suffering from neuromuscular disease
* children presenting symptoms of chronic respiratory disease before ARDS

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children hospitalised in PICU with ARDS and surviving 1 year after the acute phase
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2006-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Dynamic lung compliance | 1 year +- 2 months after discharge from ICU

SECONDARY OUTCOMES:
respiratory complaints (cough, wheeze,dypnea at rest on exertion, bronchitis, pneumonia | 1 year +- 2 months after discharge from ICU
extend of ground glass opacification (CT scan) | 1 year +- 2 months after discharge from ICU
extend of intense parenchymal opacification | 1 year +- 2 months after discharge from ICU
extend of reticular pattern | 1 year +- 2 months after discharge from ICU
extend of decreased attenuation due to emphysema | 1 year +- 2 months after discharge from ICU
extend of decreased attenuation attributable to small-airway disease | 1 year +- 2 months after discharge from ICU
carbon monoxide diffusing capacity | 1 year +- 2 months after discharge from ICU
Pulse oxymetry oxygen saturation at the end of a 6 min walk test | 1 year +- 2 months after discharge from ICU

CONTACTS AND LOCATIONS:
Overall Officials: Francis Leclerc, MD, Study Chair — University hospital of Lille , France
Locations (5):
- Hôpital Universitaire des Enfants Reine Fabiola, Université Libre de Bruxelles,, Brussels, Belgium
- France (4):
  - Hôpital Jeanne de Flandre, Centre Hospitalier Régional et Universitaire de Lille, Lille
  - Hôpital Trousseau, Assistance Publique Hôpitaux de Paris, Paris
  - Hôpital Robert Debré, Assistance Publique Hôpitaux de Paris, Paris
  - Hôpital Necker-Enfants Malades, Assistance Publique Hôpitaux de Paris, Paris

REFERENCES:
- [Derived] Neve V, Sadik A, Petyt L, Dauger S, Kheniche A, Denjean A, Leger PL, Chalard F, Boule M, Javouhey E, Reix P, Canterino I, Deken V, Matran R, Leteurtre S, Leclerc F. Whole pulmonary assessment 1 year after paediatric acute respiratory distress syndrome: prospective multicentre study. Ann Intensive Care. 2022 Aug 20;12(1):79. doi: 10.1186/s13613-022-01050-4. PMID 35986824